CLINICAL TRIAL: NCT01202331
Title: Tripartite International Research for the Elimination of Trachoma
Acronym: TIRET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Thomas M. Lietman, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-02169
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Trachoma; Chlamydia
Keywords: Bacterial Infections; Chlamydia Infections; Eye Diseases
MeSH Terms: conditions — Trachoma; Chlamydia Infections; Bacterial Infections; Eye Diseases | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- J (No Intervention): Stop Annual Treatment
- K (No Intervention): Stop Biannual Treatment
- L (Other): Continue Annual Treatment
  Interventions: Drug: mass treatment with oral azithromycin
- M (Other): Continue Biannual Treatment
  Interventions: Drug: mass treatment with oral azithromycin
- N (Experimental): Targeted Treatment by Age
  Interventions: Drug: mass treatment with oral azithromycin
- O (Experimental): Targeted Treatment by Clinical Exam
  Interventions: Drug: mass treatment with oral azithromycin

INTERVENTIONS:
Drug: mass treatment with oral azithromycin — For baseline and follow-up surveys prior to azithromycin distribution, a stratified random sample from two age groups will be chosen: 1) 60 study participants younger than 10 years old and 2) 60 study participants aged 10 years and above. Clinical examination will be performed and conjunctival swabs will be taken from all the study participants. Nasopharyngeal swabs will be collected in each community from 15 randomly selected children among the 60 participants under age 10 who were recruited for conjunctival swabbing. Then a single dose of azithromycin will be distributed according to study design: in tablet form for adults; a weight-adjusted tablet dose for children ages 8-10; and pediatric suspension for children ages 1 - 7.
  Other Names: Zithromax
  Arms: L; M; N; O

SUMMARY:
Mass antimicrobial administrations have been remarkably successful in reducing the prevalence of the ocular strains of Chlamydia that cause trachoma. Repeated distributions progressively lower the prevalence of infection, and in some cases may even result in local elimination. Mass treatments cannot be continued forever, due to concerns about cost and antibiotic resistance. The hope has been that other measures such as latrine construction and hygiene programs would prevent infection from returning. Unfortunately, no non-antibiotic measure has yet demonstrated an effect on infection.

1. We hypothesize that Chlamydial infection will return to communities when treatment ends.
2. We hypothesize that infection will be completely eliminated in all communities treated for seven years.
3. We hypothesize that identifying and treating clinically active cases among preschool aged children will delay or even prevent reemergence at a far lower cost than mass treatment of all individuals.

DETAILED DESCRIPTION:
The proposed study is a group-randomized trial to determine the frequency and treatment target of community-wide mass antibiotic treatment to eliminate trachoma. We will continue to monitor a sub-set of communities from our TANA study, in Goncha Siso Enese district of East Gojam Zone, Ethiopia. Here we evaluate how infection returns when antibiotics are discontinued, whether infection can be predictably eliminated, and whether infection can be prevented from returning with targeted treatment strategies:

Specific Aim 1. To determine whether antibiotics can be stopped after 4 years.

Specific Aim 2. To determine whether infection can be completely eliminated if mass treatments continue for seven years.

Specific Aim 3. To determine whether treatment targeted to pre-school aged children, or to households in which a pre-school aged child has clinically active trachoma, will prevent infection from returning into the community.

Specific Aim 4: To determine whether mass azithromycin distributions reduce visits to local health clinics due to all causes and infectious causes.

Specific Aim 5: To determine whether mass azithromycin distributions result in better growth metrics (weight-for-height, height-for age, weight-for-age, middle upper arm circumference) compared to no treatment.

Specific Aim 6: To determine whether under-5 mortality is lower in communities treated with mass azithromycin compared to no treatment

Specific Aim 7: To determine whether macrolide resistance in Streptococcus pneumoniae, Hameophilus influenzae, and Staphylococcus aureus is more prevalent in communities treated with biannual mass azithromycin compared to communities treated with annual mass azithromycin, and to determine whether targeted azithromycin treatments result in less macrolide resistance compared to mass azithromycin distributions.

ELIGIBILITY:
Inclusion Criteria:

* All residents residing in the state-teams which are randomly selected for this study.

Exclusion Criteria:

* Pregnant women
* Children under 6 months of age
* All those who are allergic to macrolides or azalides
* Refusal of village chief (for village inclusion), or refusal of parent or guardian (for individual inclusion)

Individuals in these three exclusion criteria will not be given the study antibiotic azithromycin, but offered the current WHO-recommended alternative treatment to azithromycin for active trachoma, which is 1% tetracycline eye ointment, to be used twice a day, topically to both eyes, for six weeks. Note that the exclusion criteria refer to the exclusion to the treatment drug, but not to the monitoring, treatment of trachoma, and examinations.

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 29000 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The average prevalence of ocular chlamydia infection in communities in an arm as determined by pooled NAAT (Nucleic Acid Amplification Test)(at 36 months versus 0 months for Aim 1, at 36 months for Aim 2 and Aim 3) | 36 months

SECONDARY OUTCOMES:
Clinical active trachoma in community, as determined by the WHO simplified grading system | 36 months
Childhood mortality (6 months -5 years of age), 6-10 years of age, and >10 years | 36 months
Macrolide resistance in pneumococcus, Haemophilus influenzae, and Staphylococcus aureus (% resistance over time, clustered by randomization unit) | 36 months
Anthropometric measurements (weight and height), as outlined by WHO child growth standards (0-5 years of age) | 3, 12, 24, and 36 months after baseline
Health clinic visits (due to all causes and due to infectious causes) in children aged 6 months-5 years, 6-10 years, and >10 years | 36 months
Prevalence of anemia (hemoglobin levels in 0-9 year olds) and the prevalence of malaria | 36 months
Clinically active trachoma in a school (all children under age 10), as determined by the WHO simplified grading system | 36 months
Cost-effectiveness of mass azithromycin administration, per infection year prevented and cost per eliminated village | 0, 12, 24, and 36 months
Estimate of chlamydial load from real-time, qPCR | 0, 12, 24, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Tom Lietman, MD, Principal Investigator — F.I. Proctor Foundation, UCSF; Kieran S O'Brien, MPH, Study Director — F.I. Proctor Foundation, UCSF; Paul Emerson, PhD, Study Director — Emory University
Locations (1):
- The Carter Center, Ethiopia, Addis Ababa, Ethiopia

REFERENCES:
- [Derived] Mahmud H, Haile BA, Tadesse Z, Gebresillasie S, Shiferaw A, Zerihun M, Liu Z, Callahan EK, Cotter SY, Varnado NE, Oldenburg CE, Porco TC, Lietman TM, Keenan JD. Targeted Mass Azithromycin Distribution for Trachoma: A Community-Randomized Trial (TANA II). Clin Infect Dis. 2023 Aug 14;77(3):388-395. doi: 10.1093/cid/ciad211. PMID 37021692
- [Derived] Keenan JD, Gebresillasie S, Stoller NE, Haile BA, Tadesse Z, Cotter SY, Ray KJ, Aiemjoy K, Porco TC, Callahan EK, Emerson PM, Lietman TM. Linear growth in preschool children treated with mass azithromycin distributions for trachoma: A cluster-randomized trial. PLoS Negl Trop Dis. 2019 Jun 5;13(6):e0007442. doi: 10.1371/journal.pntd.0007442. eCollection 2019 Jun. PMID 31166952
- [Derived] Keenan JD, Tadesse Z, Gebresillasie S, Shiferaw A, Zerihun M, Emerson PM, Callahan K, Cotter SY, Stoller NE, Porco TC, Oldenburg CE, Lietman TM. Mass azithromycin distribution for hyperendemic trachoma following a cluster-randomized trial: A continuation study of randomly reassigned subclusters (TANA II). PLoS Med. 2018 Aug 14;15(8):e1002633. doi: 10.1371/journal.pmed.1002633. eCollection 2018 Aug. PMID 30106956